CLINICAL TRIAL: NCT07045584
Title: Temporal Pole Transcranial Alternating Current Stimulation for Children With Autism Spectrum Disorder: A Randomized Controlled Open-Label Trial
Brief Title: Temporal Pole Transcranial Alternating Current Stimulation for Children With Autism Spectrum Disorder
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fei Li (Other)
Responsible Party: Sponsor-Investigator, Fei Li, Chief Physician, Doctoral Supervisor, Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Organization: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XHEC-C-2025-090-3
Record Dates: First submitted 2025-05-29; First posted 2025-07-01 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism Spectrum Disorder (ASD); Transcranial Alternating Current Stimulation (tACS); Transcranial temporal interference stimulation (tTIS); Children; Intervention
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Blinding of Clinical Scale Assessors
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention group(tACS) (Experimental): Receive tACS stimulation targeting the temporal pole, with stimulation frequency of 40Hz, using adapter power supply: voltage 9V, current set at 1.5mA, 6 times/day, 20min/session with 20min intervals between sessions, lasting for 5 days
  Interventions: Device: Transcranial Alternating Current Stimulation
- Control group (No Intervention): Receive routine rehabilitation training during the study period
- Intervention group(tTIS) (Experimental): Receive tTIS targeting the temporal pole, with stimulation frequency of 2040/2000HZ, using battery power supply: voltage 12V, current set at 1.5mA, 6 times/day, 20min/session with 20min intervals between sessions, lasting for 5 days
  Interventions: Device: transcranial Temporal Interference Stimulation

INTERVENTIONS:
Device: Transcranial Alternating Current Stimulation — Intervention Group（tACS）: Receive tACS stimulation targeting the temporal pole, with stimulation frequency of 40Hz, using adapter power supply: voltage 9V, current set at 1.5mA, 6 times/day, 20min/session with 20min intervals between sessions, lasting for 5 days;
  Arms: Intervention group(tACS)
Device: transcranial Temporal Interference Stimulation — Intervention Group（tTIS）: Receive tTIS targeting the temporal pole, with stimulation frequency of 2040/2000HZ, using battery power supply: voltage 12V, current set at 1.5mA, 6 times/day, 20min/session with 20min intervals between sessions, lasting for 5 days;
  Arms: Intervention group(tTIS)

SUMMARY:
The goal of this open-label randomized controlledl trial is to explore the safety and efficacy of conventional transcranial alternating current stimulation (tACS) and transcranial temporal interference stimulation (tTIS) targeting the temporal pole in children with autism spectrum disorder (ASD) in China. The main questions it aims to answer are:

*Can tACS and tTIS safely and effectively improve clinical symptoms in children with autism?

Researchers will compare the tACS group and tTIS group with control group to explore the safety, feasibility and efficacy of the transcranial electrical stimulation in children with autism.

Participants will:

* tACS group: undergo 5 days of temporal pole tACS
* tTIS group:undergo 5 days of temporal pole tTIS
* Control group: receive routine rehabilitation training during the study period.

From baseline to 4 weeks after intervention completion, subjects will be followed up regarding clinical symptoms and adverse reactions:

* Safety Outcome Measures: adverse events
* Primary Efficacy Outcome Measures: Social Responsiveness Scale (SRS-2) total scores
* Other clinical outcome measures related language, adapative function and cognition

DETAILED DESCRIPTION:
This research is a 5-week prospective, open-label, randomized controlled trial, planning to enroll 36 autistic children aged 4-10 with a full-scale intelligence quotient (FSIQ) of 50 or above. Children who satisfy all inclusion criteria without meeting any exclusion criteria, may be enrolled after their legal guardians provided the written informed consent.

Eligible subjects will be randomly divided into three groups: tACS group, tTIS group and control group. The tACS group will undergo 5 days of temporal pole tACS stimulation (1.5mA, 40Hz, 20min/session, 6 sessions/day); the tTIS group will undergo 5 days of temporal pole TI stimulation（1.5mA, 2040/2000Hz, 20min/session, 6 sessions/day）; the control group will receive routine rehabilitation training during the study period, including various rehabilitation services provided by the community.

At baseline, subjects will undergo physical measurements, demographic and medical history collection, intelligence test and symptom clinical scale assessments, and resting-state EEG collection. From the start of intervention until 4 weeks after completion, subjects will be followed up regarding clinical symptoms, neuroimaging, and adverse reactions.

The safety outcome: adverse events and their rate. The primary efficacy outcome is the change in Social Responsiveness Scale (SRS-2) scores 4 weeks after intervention completion compared to pre-intervention.

Secondary outcomes include changes in SRS-2 scores immediately after the 5-day intervention compared to pre-intervention; and changes in Chinese Communicative Development Inventory (CCDI), Childhood Autism Rating Scale (CARS), Peabody Picture Vocabulary Test (PPVT), Developmental Neuropsychological Assessment (NEPSY-II, including narrative memory, facial memory, theory of mind, vocabulary generation) four items, and Clinical Global Impression (CGI) scale scores 4 weeks after the 5-day intervention compared to pre-intervention.

Exploratory indicators include changes in resting-state EEG neuroimaging characteristics before intervention, immediately after the 5-day intervention, and 4 weeks after the 5-day intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged 4-10 years
2. Meeting the diagnostic criteria for ASD according to the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5)
3. Diagnosis confirmed by the Autism Diagnostic Observation Schedule (ADOS) and/or the Autism Diagnostic Interview-Revised (ADI-R)
4. Full Scale Intelligence Quotient (FSIQ) ≥50
5. Signed informed consent form

Exclusion Criteria:

1. Individuals with metal implants in the body
2. Individuals with neurological disorders such as epilepsy
3. Those requiring surgical treatment due to structural abnormalities indicated by brain MRI examination
4. Those diagnosed with genetic or chromosomal abnormalities
5. Individuals with mental illness (such as mood disorders, etc.)
6. Those with severe cardiac disease
7. Individuals with increased intracranial pressure
8. Those currently participating in other clinical trials
9. Those who received new intervention protocols within 4 weeks prior to enrollment.

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-11-20 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Social Responsiveness Scale, SRS-2 | Baseline, 4 weeks after completion of 5-day intervention
  The SRS-2 is primarily used to assess symptoms associated with ASD. Compared to other autism assessment tools, the SRS-2 stands out for its focus on quantifying the severity of social impairment, with higher scores indicating more autism symptoms and greater social disability.

SECONDARY OUTCOMES:
SRS-2 | Baseline, after completion of 5-day intervention
  The SRS-2 is primarily used to assess symptoms associated with ASD. Compared to other autism assessment tools, the SRS-2 stands out for its focus on quantifying the severity of social impairment, with higher scores indicating more autism symptoms and greater social disability.
Childhood Autism Rating Scale (CARS) | Baseline, 4 weeks after completion of 5-day intervention
  CARS is a behavior rating scale used to assess the presence and severity of the symptoms associated autism spectrum disorder. The scores of the CARS rate from 15 to 60, and higher scores indicate more severe symptoms. The changes in the CAR scores from baseline to 3 months after the treatment will be analyzed to asses the impact often intervention on participants with ASD.
Chinese Communicative Development Inventory, CCDI | Baseline, 4 weeks after completion of 5-day intervention
  Chinese Communicative Development Inventory(CCDl)is a questionnaire used to measures the language abilities. Higher scores suggest better language level. The changes in the CCDl between baseline and 3 month after treatment will be analyzed.
Peabody Picture Vocabulory Test, PPVT | Baseline, 4 weeks after completion of 5-day intervention
  PPVT as a tool for measuring children's language receptive ability and language comprehension ability
Neuropsychological Assessment for Child, NEPSY-II | Baseline, 4 weeks after completion of 5-day intervention
  NEPSY-II is a comprehensive neuropsychological measurement tool used for assessing neuro-cognitive functions in children aged 3-16 years. This study primarily evaluates four aspects: narrative memory assessment; facial memory assessment; theory of mind; and word generation.
Vineland Adaptive Behavior Scales-Third Edition, Vineland-3 | Baseline, 4 weeks after completion of 5-day intervention
  The VABS-3 is used to measure adaptive functioning across domains such as communication,daily living skills,socialization,and motor skills.Changes in VABs scores from baseline to 3 months post-treatment will be analyzed to assess the intervention's impact on adaptive behaviors in children with ASD.
Clinical Global Impression Scale (CGI) | after completion of 5-day intervention, four weeks after completion of 5-day intervention
  The Clinical Global Impressions (CGI) scale is used to assess both the severity of illness and the global improvement of participants undergoing intervention.The Clinical Global Impression-Severity scale (CGI-S) is a clinician-rated, 7-point scale that measures overall illness severity. Scores range from 1 (Normal, not at all ill) through 4 (Moderately ill) to 7 (Among the most extremely ill patients).
  The Clinical Global Impression-Improvement scale (CGI-I) is a companion measure that evaluates changes in the patient's symptoms relative to baseline. Scores range from 1 (Very much improved) through 4 (No change) to 7 (Very much worse).The CGI-E thus yields an efficacy index (EI) that reflects the net clinical benefit, accounting for both symptom improvement and adverse effects.

OTHER OUTCOMES:
Several electroencephalography (EEG) parameters | Baseline, after completion of 5-day intervention, 4 weeks after completion of 5-day intervention
  Several electroencephalography (EEG) parameters, including power spectrum and inter-trial phase coherence (ITPC) in the alpha and theta frequency bands at different time points

CONTACTS AND LOCATIONS:
Locations (1):
- Xinhua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
The study Protocol, statisticalAnalysis plan, informed Consent Form, and other relevant documents wil be available under reasonable and ethically approved request to the corresponding authors.